CLINICAL TRIAL: NCT00573521
Title: Risk Factors for Piperacillin/Tazobactam Resistance in Extended-Spectrum Beta-Lactamase (ESBL) Producing Organisms
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Brian Potoski, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO07100136
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Enterobacteriaceae Infections
Keywords: ESBL positive cultures
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This research will be conducted to determine whether risk factors exist for piperacillin/tazobactam resistance in ESBL organisms.

DETAILED DESCRIPTION:
This is chart review at UPMC. NO human subject interaction will occur.

ELIGIBILITY:
Inclusion Criteria:

* Clinical information is collected by chart review of "case" and "control" patients.
* A "case A" patient is defined as follows: One or more clinical cultures are positive for an ESBL producing bacteria and the organism is piperacillin/tazobactam resistant.
* A "case B" patient is defined as follows: One or more clinical cultures are positive for an ESBL producing bacteria and the organism is piperacillin/tazobactam susceptible.
* Additionally, 1 control patient in the hospital at the same time as the case patients will be randomly selected for each case and are not in either case group.

Exclusion Criteria:

* Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESBL positive cultures
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2007-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
This research will help to identify risk factors for resistance to an antibiotic that is commonly used in the empiric treatment of critically ill patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Potoski, Pharm D, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States